CLINICAL TRIAL: NCT01791712
Title: Enhanced Vascular Endothelial Growth Factor and Pro-inflammatory Cytokine Clearances With On-line Hemodiafiltration Versus High-flux Hemodialysis in Sepsis-related Acute Kidney Injury Patients
Brief Title: Efficacy of Online Hemodiafiltrationlysis in Cytokine Removal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Khajohn Tiranathanagul, Doctor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KJWW367/53
Record Dates: First submitted 2011-10-11; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- On-line hemodiafiltration (Experimental): On-line hemodiafiltration is a type of renal replacement therapy that was assigned as the intervention to compare with the control arm
  Interventions: Procedure: On-line hemodiafiltration
- High-flux hemodialysis (control) (Active Comparator): The standard high-flux hemodialysis is the routine renal replacement therapy in sepsis-related acute kidney injury patients and is assigned as the intervention for the control group.
  Interventions: Procedure: High-flux Hemodialysis

INTERVENTIONS:
Procedure: On-line hemodiafiltration — pre-dilution 40% of blood flow rate blood flow rate 300-350 ml/min dialysate flow rate 800 ml/min
  Other Names: Nikkiso dialysis machine; ARROW dual lumen dialysis catheter; PureFlux -150H synthetic membrane dialyzer
  Arms: On-line hemodiafiltration
Procedure: High-flux Hemodialysis — blood flow rate 300-350 ml/min dialysate flow rate 800 ml/min
  Arms: High-flux hemodialysis (control)

SUMMARY:
Following the concept of "peak concentration hypothesis", which suggest the cutting peak of pro- and anti-inflammatory mediators would result in restoring a situation of immunohomeostasis. The investigators conducted the prospective randomized controlled trial aimed to compare the clearance efficacy between on-line hemodiafiltration and high-flux hemodialysis in sepsis-related acute kidney injury patients. The lowering cytokines level during sepsis is postulated to improved outcomes in sepsis.

DETAILED DESCRIPTION:
1. Blood samples were taken from patients before and at the end of 4-hour in the first dialysis session. The percentage of reductions were calculated from the before and ending samples. The values of postfilter samples were corrected for changes in plasma volume, based on hemoglobin (Hb) of prefilter.
2. VEGF and other cytokines (IL-6, IL-8, IL-10, and TNF-α) were determined in the plasma separated from EDTA blood. After collection, plasma separation was achieved by centrifugation for 10 min at 1,500 g. Immediately after separation, the samples were stored at -70 ºC until further analysis.
3. All determinations were carried out in duplicate. The panels of cytokines (VEGF, IL-6, IL-8, IL-10, and TNF-α) were measured using the Luminex xMap-based multiplex technology. Assays were performed using the MILLIPLEX MAP (multi-analyte panels) 5-plex Cytokine Kit (Millipore, Billerica, MA) on the Luminex® instrument according to the manufacturer's procedure.

ELIGIBILITY:
Inclusion Criteria:

* Sepsis
* acute kidney injury (RIFLE classification F)
* Age more than 18

Exclusion Criteria:

* Hemodynamic instability
* Whom written informed consent could not be obtained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Reduction in plasma Vascular Endothelial Growth Factor (VEGF)level | At time 0-hour and 4-hour of the study dialysis session

SECONDARY OUTCOMES:
Intradialytic hypotension | During 4 hours of the study dialysis session
Renal recovery (at 30 days) | participants will be followed for the renal recovery (dialysis-free) for the 30 days from the first initiation of dialysis
Hospital patient mortality | participants will be followed for the duration of hospital stay (an expected average of 5 weeks)
  mortality during hospital admission

CONTACTS AND LOCATIONS:
Overall Officials: Khajohn Tiranathanagul, M.D., Principal Investigator — Chulalongkorn University; Wiwat Chancharoenthana, M.D., Principal Investigator — Chulalongkorn University
Locations (1):
- King Chulalongkorn Memorial Hospital, Bangkok, Bangkok, Thailand